CLINICAL TRIAL: NCT05735418
Title: A Study on the Effects of Oral Intake of GI Biome #7 on the Intestinal Microbiome and Health in the Elderly Population
Brief Title: The Effect of GI Biome #7 on Gut Microbiome and Health of the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: GI Biome (Unknown)
Responsible Party: Principal Investigator, Yun-Chul Hong, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIB-2022-088
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Muscle Weakness
Keywords: gut microbiome; probiotics; muscle strength; intervention
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: A double-blind, randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GI Biome #7 (Experimental): The intervention consists of daily administration of probiotics GI Biome #7 for four weeks.
  Interventions: Dietary Supplement: GI Biome #7
- Placebo (Placebo Comparator): The placebo consists of daily administration of the placebo pills made up of 100% maltodextrin for four weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: GI Biome #7 — It comprises probiotics (Lactobacillus fermentum, Lactobacillus acidophilus, Lactobacillus plantarum, and Bifidobacterium animalis ssp. lactis) and prebiotics (vitamin B2., Korean red ginseng, and etc.). The administration dosage of probiotics is 5×10^8 CFU/day.
  Arms: GI Biome #7
Dietary Supplement: Placebo — The placebo consists of daily administration of the placebo pills made up of 100% maltodextrin for four weeks.
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of probiotics named GI Biome #7 on the gut microbiome and muscle strength in older adults aged 60 years or older.

DETAILED DESCRIPTION:
This study is a double-blind, randomized controlled trial. A total of 60 healthy adults aged 60 years or older will be recruited, and they will be randomly assigned to the intervention group or the control group. The intervention group will be given GI Biome #7 pills, and the control group will be given the placebo pills for four weeks. The participants will visit the research laboratory four times as follows: A day before starting to take the pills, two weeks later after starting to take the pills, the last day of taking the pills, and four weeks later after the end of taking the pills. Participants' stool, blood, and urine will be sampled every visit, and grip strength and body composition will also be checked.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or older
* Those who have no difficulties in daily living
* Willing to commit throughout the study

Exclusion Criteria:

* Antibiotics medication in the last month.
* Probiotics used in the last months.
* Those who are in the treatment of the following diseases: Liver disease, Neurological disease, Respiratory disease, Tumors, Psychiatric disorders, Angina, Myocardial infarction, and Stroke

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Hand Grip Strength Change | 4 weeks
  Change from baseline hand grip strength at 4 weeks

SECONDARY OUTCOMES:
Bacteroidetes/Firmicutes Ratio Change | 4 weeks
  Change from baseline Bacteroidetes/Firmicutes ratio in gut microbiome at 4 weeks
Fasting blood glucose | 4 weeks
  Change from baseline fasting blood glucose at 4 weeks

OTHER OUTCOMES:
Walking speed | 0, 2, 4, 8 weeks
  The time to walk a 10-m distance will be measured.
Gut quotient | 0, 2, 4, 8 weeks
  Gut quotient measurement scales will be asked using questionnaires. The minimum and maximum values are 0 and 100, respectively. Higher scores are related to worse gut quotient.
IGF-1 | 0, 2, 4, 8 weeks
  IGF-1 will be quantified from the participants' serum samples.
Myostatin | 0, 2, 4, 8 weeks
  Myostatin will be quantified from the participants' serum samples.
8-OHdG | 0, 2, 4, 8 weeks
  8-OHdG will be quantified from the participants' serum samples.
Fecal acetate level | 0, 2, 4, 8 weeks
  Acetate level (short-chain fatty acid) will be measured from the participants' stool.
Fecal butyrate level | 0, 2, 4, 8 weeks
  Butyrate level (short-chain fatty acid) will be measured from the participants' stool.
Fecal propionate level | 0, 2, 4, 8 weeks
  Propionate level (short-chain fatty acid) will be measured from the participants' stool.
Fecal calproate level | 0, 2, 4, 8 weeks
  Calproate level (short-chain fatty acid) will be measured from the participants' stool.
Fecal valerate level | 0, 2, 4, 8 weeks
  Valerate level (short-chain fatty acid) will be measured from the participants' stool.

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Chul Hong, MD, PhD, Study Director — Seoul National University
Locations (1):
- Seoul National University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No